CLINICAL TRIAL: NCT05398770
Title: Randomized Clinical Trial on the Effect of Vitamin D Supplement Prior to Non-surgical Periodontal Therapy: a Feasibility Trial
Brief Title: Vitamin D Supplementation Prior to Non-surgical Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: Public Dental Service Competence Center of Northern Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2022/440018
Record Dates: First submitted 2022-05-25; First posted 2022-06-01 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis; Periodontal Diseases; Periodontal Inflammation; Inflammation; Inflammation Gum; Vitamin D
Keywords: Vitamin D; 25(OH)D; Cholecalciferol; Periodontitis
MeSH Terms: conditions — Periodontitis; Periodontal Diseases; Inflammation; Gingivitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin D3 (30 µg/d) (Experimental): Subjects will take 30 µg vitamin D3 per day
  Interventions: Dietary Supplement: Vitamin D supplementation (30 µg/d)
- Placebo (Placebo Comparator): Subjects will take placebo
  Interventions: Dietary Supplement: Vitamin D supplementation (30 µg/d)

INTERVENTIONS:
Dietary Supplement: Vitamin D supplementation (30 µg/d) — The participants will be instructed to take the tablets (vitamin D or placebo) once a day 4 weeks prior to the onset of the non-surgical periodontal treatment (NSPT), and to continue for two weeks after their first NSPT, altogether 6 weeks.

SUMMARY:
The purpose of this study is to test the feasibility i. e. to examine all aspects necessary for the implementation of a future randomized clinical trial (RCT) that aims to determine whether non-surgical periodontal treatment can be improved by concomitant intake of vitamin D.

DETAILED DESCRIPTION:
Vitamin D is believed to have anti-inflammatory and anti-bacterial properties. This is hypnotized to play a role in periodontitis. Well-designed RCTs on this theme are lacking. We therefore aim at testing a proposed study design in a pilot study, on vitamin D supplementation and its possible adjunctive effect on non-surgical periodontitis treatment (NSPT).

Altogether 28 patients with a referral for treatment at the Public Dental Service Competence Center of Northern Norway (TkNN), diagnosed with periodontitis Stage I-IV, and within the ages of 20-60 years will be recruited. Participation is voluntary and based on written informed consent.

The participants will randomly be allocated into two groups of equal sizes. The intervention group will receive vitamin D supplementation of 30 µg/day, and the control group will receive placebo tablets. The study is double-blinded.

The participants will be instructed to take the tablets once a day for four weeks prior to the onset of the NSPT, and for two additional weeks after their first NSPT, altogether six weeks. The aim is to ensure that the vitamin D status among those who receive vitamin D supplementation is satisfactory at the start of NSPT and throughout the NSPT period.

At baseline and before the start of intervention a dentist will perform a periodontal examination, including bleeding on probing (BoP), probing pocket depth (PPD), determine lost teeth, mobility, furcation involvement and radiographic bone loss. Clinical measurements in addition to data on age and sex will be obtained from the clinics (TkNN) own medical record system. The participants will also be asked to fill out a digital questionnaire about weight and height, oral hygiene, oral health, and general health. The questions in the questionnaire will be repeated at the end of follow-up, in addition to questions on the whether or not the participants have taken the tablets as prescribed, their experienced in doing so, and finally on behaviors that affect vitamin D status (taken other supplements / use of solarium / sun holidays).

At baseline, at week five and at the end of the study period, gingival crevicular fluid (GCF) and blood samples from blood vessels in the arm will be sampled and analyzed for their content of vitamin D, inflammatory markers and enzymes. As a secondary outcome we also aim to assess the correlations between levels of inflammatory markers in blood and the GCF.

The duration of follow-up depends on how many treatments the dentist considers the patient will need. This is part of the ordinary treatment regimen offered to this patient group. The treatment will take place over a time-period of one month. The patient is then invited to return for a check-up after 6-8 weeks. The total estimated time that each individual will be involved in the study is approximately 11-13 weeks.

Once the pilot study is completed, all steps (both scientific and practical) of the trial will be evaluated in details to assess what worked / did not work / could have worked better - including recruitment, randomization, follow-up, dropout, reason for dropout, patient compliance, side effects, GCF and blood samples; including sampling storage, shipping, analysis and more.

The benefits of running a feasibility trial is that it provides valuable insight and knowledge useful for designing and conducting a future high quality clinical trial on this topic. If vitamin D is confirmed to improve the effect of NSPT in a future clinical trial, improving vitamin D status in patients would be an easy to carry out means in the fight against this disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic periodontitis according to the 2017 case definition
* Adults, age group 20-60 years
* Periodontitis Stage I-IV (2017 definition)

Exclusion Criteria:

* Systemic illnesses (diabetes, osteoporosis)
* Smoking
* Immuno-suppressive treatment
* Pregnancy
* Daily vit-D supplements
* Solarium
* NSPT within 6 months
* Local anti-microbial treatment
* No natural teeth/peri implantitis

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Change in periodontitis status after treatment (2017 case definition) | Changes from baseline at week 5
  Bleeding on probing (BOP)
Change in periodontitis status after treatment (2017 case definition) | Changes from week 5 to week 11-13
  Bleeding on probing (BOP)
Change in periodontitis status after treatment (2017 case definition) | Changes from baseline at week 11-13
  Bleeding on probing (BOP)
Change in periodontitis status after treatment (2017 case definition) | Changes from baseline at week 5
  Probing pocket depths (PPD)
Change in periodontitis status after treatment (2017 case definition) | Changes from week 5 to week 11-13
  Probing pocket depths (PPD)
Change in periodontitis status after treatment (2017 case definition) | Changes from baseline at week 11-13
  Probing pocket depths (PPD)

SECONDARY OUTCOMES:
Change in 25(OH)D after intervention | Changes from baseline at week 5
  Plasma concentration of 25(OH)D
Change in 25(OH)D after intervention | Changes from week 5 to week 11-13
  Plasma concentration of 25(OH)D
Change in 25(OH)D after intervention | Changes from baseline at week 11-13
  Plasma concentration of 25(OH)D
Change in biomarkers (IL-1β, IL-6, IL-8, IL-12, TNFα, CRP, MCP-1, MMP) over time as response to the intervention | Changes from baseline at week 5
  Plasma and gingival crevicular fluid concentration of biomarkers (IL-1β, IL-6, IL-8, IL-12, TNFα, CRP, MCP-1, MMP)
Change in biomarkers (IL-1β, IL-6, IL-8, IL-12, TNFα, CRP, MCP-1, MMP) over time as response to the intervention | Changes from week 5 to week 11-13
  Plasma- and gingival crevicular fluid concentration of biomarkers (IL-1β, IL-6, IL-8, IL-12, TNFα, CRP, MCP-1, MMP)
Change in biomarkers (IL-1β, IL-6, IL-8, IL-12, TNFα, CRP, MCP-1, MMP) over time as response to the intervention | Changes from baseline at week 11-13
  Plasma- and gingival crevicular fluid concentration of biomarkers (IL-1β, IL-6, IL-8, IL-12, TNFα, CRP, MCP-1, MMP)
Change in anti-microbial peptides (LL-37, hBD-2) after intervention | Changes from baseline at week 5
  Gingival crevicular fluid concentration of anti-microbial peptides (LL-37 and hBD-2)
Change in anti-microbial peptides (LL-37, hBD-2) after intervention | Changes from week 5 to week 11-13
  Gingival crevicular fluid concentration of anti-microbial peptides (LL-37 and hBD-2)
Change in anti-microbial peptides (LL-37, hBD-2) after intervention | Changes from baseline at week 11-13
  Gingival crevicular fluid concentration of anti-microbial peptides (LL-37 and hBD-2)

OTHER OUTCOMES:
Correlations with biomarkers in blood compared to levels in gingival crevicular fluid | Correlation at baseline
  Biomarkers in blood and gingival crevicular fluid (IL-1β, IL-6, IL-8, IL-12, TNFα, CRP, MCP-1, MMP, LL-37, hBD-2)
Correlations with biomarkers in blood compared to levels in gingival crevicular fluid | Correlation at week 5
  Biomarkers in blood and gingival crevicular fluid (IL-1β, IL-6, IL-8, IL-12, TNFα, CRP, MCP-1, MMP, LL-37, hBD-2)
Correlations with biomarkers in blood compared to levels in gingival crevicular fluid | Correlation at week 11-13
  Biomarkers in blood and gingival crevicular fluid (IL-1β, IL-6, IL-8, IL-12, TNFα, CRP, MCP-1, MMP, LL-37, hBD-2)
Change in self-reported oral health before and after treatment | Changes from baseline at end of follow-up (week 11-13)
  Self-reported oral health (questionnaire 5 point scale 1=bad, 5=very good)
Change in self-reported general health before and after treatment | Changes from baseline at end of follow-up (week 11-13)
  Self-reported general health (questionnaire 5 point scale 1=bad, 5=very good)

CONTACTS AND LOCATIONS:
Overall Officials: Magritt Brustad, Dr. Scient, Principal Investigator — Department of Community Medicine, University of Tromso
Locations (1):
- Public Dental Service Competence Centre of Northern Norway, Tromsø, Postboks 2406, Norway

IPD SHARING:
Plan to Share IPD: No